CLINICAL TRIAL: NCT04398472
Title: Evaluation of the Nextdoor KIND Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swinburne University of Technology (Other)
Collaborators: Brigham Young University (Other); University of Sydney (Other); University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ND01
Record Dates: First submitted 2020-03-04; First posted 2020-05-21 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Loneliness; Social Isolation
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Challenge (Active Comparator): Participants in the challenge will be asked to complete four activities over the next four weeks to address loneliness and social isolation in their communities.
  The activities will involve doing an activity with people in their neighbourhood. These activities have been selected based on being positive, engaging and feasible to the average individuals. An example of the type of activities is having a conversation with a neighbour on the phone or via video chat and safely checking in on someone who is elderly or living alone. All activities will adhere to the relevant country or states health department's safety recommendations and laws during COVID-19.
  Hypothesis 1 (H1). There will be a reduction in the primary outcome, loneliness in participants assigned to the Nextdoor KIND Challenge groups compared to the waitlist control group post the 4-week intervention
  Interventions: Behavioral: KIND Challenge
- Waitlist (No Intervention)

INTERVENTIONS:
Behavioral: KIND Challenge — The KIND challenge consists of nominating an activity to complete over a 4 week period. The activities involve doing an activity with others in your neighbourhood. These activities are positive, engaging and feasible to the average individual. Activities adhere to relevant country or state department health and safety guidelines. For example; having a chat with a neighbour online, or bringing in rubbish bins for an elderly neighbour.
  Arms: Challenge

SUMMARY:
There is ample evidence showing that loneliness is a public health problem that influences social, mental and physical health. The current project is about evaluating the effectiveness of the Kindness Is NextDoor (KIND) Challenge, a social networking platform aimed at reducing loneliness and social isolation in specific Nextdoor communities within Australia. As the landscape through which people make social connections changes due to technology it is important to evaluate the effectiveness of platforms that are designed to reduce loneliness within communities. This is the first study of its kind in Australia and will help provide insight into how to target social isolation and loneliness within communities using social networking platforms.

ELIGIBILITY:
Inclusion Criteria:

* Community dwellers who use the Nextdoor platform.
* Aged 18 to 90 years old.

Exclusion Criteria:

- Individual's without proficient English reading comprehension skills will be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4500 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Change in loneliness as measured by UCLA Loneliness Scale - Version 3 (UCLA-LS; Russell, 1996). | Challenge: 3 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, Waitlist: 4 times points: baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  The UCLA-LS is a 20-item measure employing a 1 (Never) to 4 (Always) Likert-type scale. The measure consists of both positively- and negatively-worded items that assess loneliness (e.g., How often do you feel that you are no longer close to anyone?). The UCLA-LS has been shown to correlate negatively with life satisfaction and perceived social support, thus supporting its convergent validity with related constructs. The range of possible scores is from 0-80 where higher scores indicate higher levels of loneliness.

SECONDARY OUTCOMES:
Change in quality of life as measured by European Health Interview Survey-Quality Of Life - 8-Item Index (EUROHIS-QOL-8; Power, 2003; Schmidt, Mühlan, & Power, 2005). | Challenge: 3 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, Waitlist: 4 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  The EUROHIS-QOL-8 is an 8-item measure of quality of life consisting of questions that assess overall QOL, general health, energy, daily living activity, self-esteem, social relationships, finances and home. The measure is derived from the WHOQOL-BREF and shares a similar 5-point Likert-scale response format. The scale has demonstrated good qualities in term of internal consistency (Cronbach's alpha = 0.83) and satisfactory convergent and discriminant validity (Schmidt et al., 2005). The range of possible scores is 8-40 where higher scores indicate higher quality of life.
Change in depression as measured by Patient Health Questionnaire-8 (PHQ-8; Kroenke & Spitzer, 2002). | Challenge: 3 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, Waitlist: 4 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  The PHQ-8 is an 8-item measure of depression severity based on 8 of the 9 item criteria of the DSM-IV. The measure was derived from the PHQ-9 however; the ninth question was omitted from this study as depression was not a primary outcome. Depression severity is scored based on the presence of depressive symptomology in the previous 2 weeks of measure admission. The scale uses a 1 (not at all) to 4 (nearly every day) Likert scale with higher scores indicating higher levels of depressive symptomology. The range of possible scores is 8-32. The PHQ-9 has been shown to have good criterion and construct validity and excellent internal consistency (Kroenke, Spitzer, & Williams, 2001). The PHQ-8 shares similar properties in terms of validity and reliability and is therefore an adequate alternative to its 9-item scale counterpart (Kroenke & Spitzer, 2002).
Change in social anxiety as measured by Mini-Social Phobia Inventory (Mini-SPIN; Connor, Kobak, Churchill, Katzelnick, & Davidson, 2001). | Challenge: 3 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, Waitlist: 4 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  The Mini-SPIN is a brief 3-item measure of generalised social anxiety disorder. The measure employs a 5-point Likert scale form 1 (not at all) to 5 (extremely), with higher scores indicating a greater level of generalised social anxiety. The range of possible scores is 3-15. The Mini-SPIN has shown high sensitivity in detecting social anxiety disorder (Connor et al., 2001).
Change in perceived stress as measured by Perceived Stress Scale-4 (PSS-4; Cohen, Williamson, Spacapan, & Oskamp, 1988). | Challenge: 3 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, Waitlist: 4 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  This four-item measure of stress was derived from the original 14-item Perceived Stress Scale (PSS). This measure consists of both positively and negatively worded items that asses an individual's evaluation of stressful events. The measure employs a 5-point Likert scale ranging from 0 (never) to 4 (very often). The range of possible scores is 0-16 where higher scores indicate higher levels of perceived stress. The PSS-4 has been shown to negatively correlate with levels of perceived health, social support, being male, and older age (Warttig, Forshaw, South, & White, 2013). The scale has demonstrated fair reliability and adequate psychometric properties (Warttig et al., 2013).
Change in positive and negative affect as measured by The Positive and Negative Affect Schedule-Short Form (PANAS-SF 10 item; Watson, Clark, & Tellegen, 1988) | Challenge: 3 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, Waitlist: 4 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  The PANAS-SF is a 10-item short form version of the Positive and Negative Affect Scale scale. The measure asks respondents to rate the extent to which they feel a particular emotion along a 5-point Likert scale ranging from 1 (very slightly) to 5 (extremely). The range of possible scores is 5-25 for each subscale (positive affect and negative affect) where higher scores indicate higher levels of positive or negative affect. This subscale measure has been shown to have high levels of internal consistency (Watson et al., 1988) and acceptable levels of convergent validity (Roesch, 1998).
Change in social cohesion and community trust as measured by the Social Capital Scale (Martin, Rogers, Cook, & Joseph, 2004). | Challenge: 3 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, Waitlist: 4 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  The Social Capital Scale is a 7-item measure designed to assess social cohesion and trust in a community. The scale was derived from a similar scale used in Sampson, Raudenbush, and Earls (1997). This measure consists of both positively and negatively worded items and is recorded on a 2 point Likert scale ranging form 0 (strongly disagree or disagree) to 1 (strongly Agree or agree). The range of possible scores is 0-14 where higher scores indicate higher levels of social cohesion and trust. This measure was shown to be a reliable tool to measure social cohesion and trust at a neighbourhood level (Sampson et al., 1997).
Neighbourhood perception of change | Challenge: 3 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, Waitlist: 4 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  This question asks if participants thought their neighbourhood was improving from 1 (improving) to 3 (declining).
Neighbourhood importance | Challenge: 3 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, Waitlist: 4 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  This question asks how important participants thought it was to know their neighbours from 1 (very important) to 5 (very important)
Neighbourhood modified Social Relationship Index | Challenge: 3 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, Waitlist: 4 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  The 3-item scale was modified from the Social Relationship Index (34). Three factors measuring support, ambivalence, and aversive. We ask how participants feel towards their neighbours when needing advice, understanding, or a favour - helpfulness, upsetting, mixed/conflicted feelings on a Likert scale from 1 (not at all) to 6 (extremely).
Neighbourhood conflict | Challenge: 3 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, Waitlist: 4 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  Participants will be asked to reflect on their interactions with their neighbours in the past month using a dichotomous yes/no to the following: absence/presence of neighbour conflict, critical comments towards the participant, participant critical of neighbours.
Neighbourhood number of contacts | Challenge: 3 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, Waitlist: 4 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  This item asks the number of people the participants knows in their neighbourhood, 0 (0-5 neighbours) to 4 (15+ neighbours).
Acceptability | 4 weeks for challenge condition, 8 weeks for waitlist
  We measured acceptability around these factors, including how connected (1 not at all connected to 10 very connected), how meaningful was the activity (1 not very meaningful to 10 very meaningful), how safe they felt when completing the challenge (1 not very safe to 10 very safe), how positive they felt (1 not very positive to 10 very positive), how comfortable they felt doing the activity (1 not at all comfortable to 10 very comfortable). It is anticipated that the Nextdoor KIND challenge will yield ratings of more than 5 indicating higher levels of acceptability across these outcomes.
Feasibility of the Challenge | 4 weeks for challenge condition, 8 weeks for waitlist
  Feasibility will be assessed by a high retention rate (i.e., <40% drop-out).
Change in social isolation risk as measured by Lubben Social Network Scale (LSNS; Lubben & Gironda, 2003). | Challenge: 3 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, Waitlist: 4 data points - baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  The LSNS is an 18-item scale that assesses the frequency and quality of contact - such as talking about private matters - in an individual's network. There are three subscales and each consists of 6 items relating to family, neighbour and friend connections. The scale employs a 0 (none) to 5 (nine or more) Likert scale and includes 6 items (eg. How many relatives do you see or hear from at least once a month?). Higher scores indicate larger social networks and lower risk of social isolation. The scale has demonstrated adequate levels of reliability and the proposed clinical cut-points showed good convergent validity (Lubben & Gironda, 2003). The range of possible scores is from 0-90 where higher scores indicate more social connections and lower risk of social isolation.
Safety of the KIND Challenge | Challenge: 4 weeks from baseline Waitlist: 8 weeks from baseline
  We assess for unintended harms (e.g., conflict) during this period. In this case, we measure the occurrence of neighbour conflict with a single dichotomous item, 'Did you have a conflict with a neighbour because of the KIND challenge'. This item is measured with a yes or no response.

CONTACTS AND LOCATIONS:
Locations (1):
- Swinburne University of Technology, Hawthorn, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim MH, Hennessey A, Qualter P, Smith BJ, Thurston L, Eres R, Holt-Lunstad J. The KIND Challenge community intervention to reduce loneliness and social isolation, improve mental health, and neighbourhood relationships: an international randomized controlled trial. Soc Psychiatry Psychiatr Epidemiol. 2025 Apr;60(4):931-942. doi: 10.1007/s00127-024-02740-z. Epub 2024 Aug 19. PMID 39158741
- [Derived] Lim MH, Qualter P, Hennessey A, Smith BJ, Argent T, Holt-Lunstad J. A randomised controlled trial of the Nextdoor Kind Challenge: a study protocol. BMC Public Health. 2021 Aug 5;21(1):1510. doi: 10.1186/s12889-021-11489-y. PMID 34353299